CLINICAL TRIAL: NCT05407181
Title: Lymphocyte Count and High Fluorescent Count (HFLC)Correlate With Liver Disorder in Dengue Fever Patients
Brief Title: Lymphocyte Count and High Fluorescent Count (HFLC) Correlate With Liver Disorder in Dengue Fever Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nurhasan Agung Prabowo (Other)
Responsible Party: Sponsor-Investigator, Nurhasan Agung Prabowo, dr. Nurhasan Agung Prabowo, Sp.PD, Universitas Sebelas Maret
Organization: Universitas Sebelas Maret (Other)
Other Study IDs: DHFandHFLC
Record Dates: First submitted 2022-06-01; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Dengue Fever
MeSH Terms: conditions — Dengue | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood and Liver Function test — Data was collected through routine blood and liver function tests using a hematology analyzer and ELISA, respectively.

SUMMARY:
Liver dysfunction marked by elevated alanine transaminase enzymes is quite common in dengue patients and subsequently affects the disease's severity and healing process. Unfortunately, liver function tests cannot always be done, especially in hospitals with limited facilities. In contrast, routine hematology tests are considered regular and inexpensive tests that can be performed on dengue patients. Therefore, this study aims to determine hematological parameters as markers of elevated liver enzymes in dengue patients.

DETAILED DESCRIPTION:
This cross-sectional study involves 11 dengue fever patients, consisting of 9 men and two women, at Sebelas Maret University Hospital (RS UNS), Sukoharjo. The study was conducted in May 2021. Inclusion criteria included patients who were hospitalised at UNS Hospital with the following criteria: (1) adult patients (19-65 years); (2) diagnosed with dengue hemorrhagic fever according to WHO 2011 criteria; (3) routine blood examination at least once in seven days since the onset of fever; and (4) checked alanine transaminase and aspartate transaminase levels at least once in seven days from the onset of fever. The research was approved by the Regional General Hospital Health Research Ethics Commission (RSUD) by Dr Moewardi Surakarta with the number 938/X/HREC/2021.

Dengue infection is classified according to WHO 2011 criteria, including dengue fever, dengue hemorrhagic fever, and dengue shock syndrome. Dengue fever has criteria in the form of acute fever with two or more other symptoms (headache, retroorbital pain, myalgia, arthralgia, rash, bleeding manifestations); laboratory investigations support dengue fever (platelets 150,000/mm3, leukocytes <5000/mm3, an increase in hematocrit 5-10%), with other confirmed assays (dengue virus isolation; fourfold increase in dengue-specific IgG or IgM serum; antigen or virus detection by immunohistochemistry, immunoassay, and ELISA; genome detection by RT-PCR). Dengue hemorrhagic fever has symptomatic criteria such as dengue fever plus signs and symptoms of plasma leakage (platelets 100,000/mm3, hematocrit increase 20%, pleural effusion, ascites, hypoproteinemia, or hypoalbuminemia). Meanwhile, dengue shock syndrome has symptomatic criteria such as dengue hemorrhagic fever plus symptoms of tachycardia and cold extremities.

Lymphocyte and HFLC examinations were carried out through a haematology analyser's routine blood tests. Meanwhile, liver function tests in aspartate transaminase and alanine transaminase were performed using ELISA. The range of normal cut-off values for each parameter is 11.7-16.2 mg/dL for hemoglobin, 35-45% for hematocrit, 3.9-5.3 x 106/mm3 for erythrocytes, 4.5-11 x 103/mm3 for leukocytes, 150-450 x 103 /mm3 for platelets, 0.8-5 x 103/mm3 for lymphocytes, 1-1.3 for NLR, and 0-1.4 for HFLC.

Data are presented using descriptive statistics and analysed using IBM SPSS (Statistical Package for the Social Sciences) Statistics 25 for Windows 10. Continuous variables are displayed using mean ± SD or median (IQR). Chi-Square tested the relationship between sex data categorical variables. The relationship between continuous variables of haematological parameter data and alanine transaminase status was tested using an unpaired t-test for normally distributed data, a Mann-Whitney test for data that were not normally distributed, and a correlation test in the form of simple logistic regression. The relationship between variables is significant if the p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients who were hospitalized at UNS Hospital with the following criteria: (1) adult patients (19-65 years); (2) diagnosed with dengue hemorrhagic fever according to WHO 2011 criteria; (3) routine blood examination at least once in seven days since the onset of fever; and (4) checked alanine transaminase and aspartate transaminase levels at least once in seven days from the onset of fever.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a cross-sectional study involving 11 dengue fever patients, consisting of 9 men and 2 women at Sebelas Maret University Hospital (RS UNS), Sukoharjo.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Estimated)
Dates: Start 2022-06-03 (Estimated); Primary Completion 2022-06-03 (Estimated); Study Completion 2022-06-05 (Estimated)

PRIMARY OUTCOMES:
Correlation of SGPT/ALT with Lymphocytes | May 30-June 5 2022
  Correlation of SGPT/ALT with Lymphocytes
Correlation of SGPT/ALT with HFLC | May 30-June 5 2022
  Correlation of SGPT/ALT with HFLC

CONTACTS AND LOCATIONS:
Overall Officials: Nurhasan Agung Prabowo, MD, Principal Investigator — Universitas Sebelas Maret
Locations (2):
- Indonesia (2):
  - RS UNS (Universitas Sebelas Maret Hospital), Sukoharjo, Central Java
  - Universitas Sebelas Maret Hospital, Sukoharjo, Central Java

IPD SHARING:
Plan to Share IPD: No